CLINICAL TRIAL: NCT03461302
Title: A Randomized Controlled Pilot Study Comparing the Efficacy of Topical Coal Tar to Topical Corticosteroids in Children Aged 1 to < 16 Years With Moderate-severe Atopic Dermatitis
Brief Title: Efficacy of Topical Coal Tar in Children With Atopic Dermatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL59682.091.16
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Coal Tar; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Coal Tar treatment (Experimental)
  Interventions: Drug: Topical coal tar
- Topical Corticosteroids treatment (Active Comparator)
  Interventions: Drug: Topical corticosteroids

INTERVENTIONS:
Drug: Topical coal tar — Solution carbonis detergens 10% in cremor vaselini lanette FNA and pix lihantracis 3% in zinc oxide paste
  Arms: Topical Coal Tar treatment
Drug: Topical corticosteroids — Clobetasone butyrate 0.05% ointment
  Arms: Topical Corticosteroids treatment

SUMMARY:
Rationale/hypothesis: Atopic dermatitis (AD) is an inflammatory skin disease, occurring most frequently in children. Currently, topically applied corticosteroids are used as a standard anti-inflammatory treatment. When a corticosteroid with a high potency is used for a long period of time, adverse effects like skin atrophy and systemic effects may occur, especially in children. In addition, corticophobia among patients is an issue that warrants alternatives for the treatment of AD in children. An alternative treatment is the topical application of coal tar, which is known to be an effective and safe treatment for AD for ages, and is used in our department for decennia. Although there is convincing evidence in the literature on the safety of coal tar, evidence in the literature on the efficacy of coal tar in the treatment of AD is lacking, especially in children.

Objective: To evaluate efficacy of topical treatment with coal tar compared to topical treatment with corticosteroids in children aged 1 to <16 years with moderate to severe AD

Study design: investigator-initiated, parallel-group randomized controlled pilot study

Study population: Children aged 1 to <16 years with moderate-severe AD

Intervention: Patients will be randomized in two groups: (1) topical treatment with coal tar or (2) topical treatment with moderate potency corticosteroids for a treatment duration of 4 weeks.

Main study parameters/endpoints: The primary outcome is the percentage change in EASI score at week 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD based on the criteria of Hanifin and Rajka
* Moderate to severe AD based on EASI score >7.1
* Willing and able to comply with visits and study-related procedures
* Provide signed informed consent (if patient >12 years of age) and/or signed informed consent provided by the parents or legal guardian (all participating patients)
* Able to understand and complete study-related questionnaires, or parent or legal guardian is able to understand and complete study-related questionnaires
* Willing to avoid excessive sunlight

Exclusion Criteria:

* Hypersensitivity and/or intolerance to topical corticosteroids or topical coal tar
* Treatment with any of the following before baseline:

  * Topical treatment with corticosteroids within 24 hours before baseline
  * Topical treatment with coal tar, tacrolimus and/or pimecrolimus within 2 weeks before baseline
  * Topical treatment with antibiotics or antifungal treatment within 7 days before baseline
  * Systemic corticosteroids, immunosuppressive/immunomodulatory drugs or phototherapy for AD within 8 weeks before baseline
  * Investigational drugs within 8 weeks or 5 half-lives (whichever is longer)
  * Use of systemic antibiotic therapy, systemic antifungal therapy and/or biologicals within 6 months before baseline
* Planned or anticipated use of any prohibited medication during the treatment and follow-up period:

  * Other medication than the prescribed study medication used for the treatment of AD, including topical calcineurin inhibitors, prescription moisturizers containing additives such as urea, antihistamines, phototherapy, systemic treatment with an immunosuppressive/immunomodulatory agent such as cyclosporine, methotrexate or biologics
  * Systemic antibiotic and/or antifungal therapy
* Indication for systemic therapy or a medical need to use a higher level of topical corticosteroids than moderate potency topical corticosteroids
* Pregnancy or breast feeding, or planning to become pregnant or breast feed
* Presence of skin co-morbidities that may interfere with study assessments
* Presence of concomitant illness that would, in the investigator's judgment, adversely affect the patient's participation in the study
* Presence of chronic hepatic or renal insufficiency
* Presence of immunodeficiency syndromes including HIV
* Presence of HBV or HCV
* Any other medical or psychological condition that would represent an unreasonable risk to the patient, make the patient's participation unreliable or interfere with study assessments

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease activity | 4 weeks
  Disease-activity measured by Eczema Area and Severity Index (EASI)

SECONDARY OUTCOMES:
Pruritus | 4 weeks
  VAS pruritus
Health-related quality of life | 4 weeks
  DLQI

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Nijmegen, Netherlands